CLINICAL TRIAL: NCT01353703
Title: Immunogenicity and Safety Study of GlaxoSmithKline Biologicals' Infanrix Hexa™ Vaccine in Healthy Infants in India
Brief Title: Immunogenicity and Safety Study in Infants of GlaxoSmithKline Biologicals' Infanrix Hexa™ (DTPa-HBV-IPV/Hib) Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 111157; 2013-003427-10 (EudraCT Number)
Record Dates: First submitted 2011-05-12; First posted 2011-05-16 (Estimated); Results first posted 2019-01-25 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Poliomyelitis; Tetanus; Acellular Pertussis; Haemophilus Influenzae Type b; Diphtheria; Hepatitis B; Diphtheria-Tetanus-aPertussis-Hepatitis B-Poliomyelitis-Haemophilus Influenzae Type b Vaccines
Keywords: Infanrix hexa™; Primary vaccination; India; combination vaccine; infants
MeSH Terms: conditions — Poliomyelitis; Tetanus; Haemophilus Infections; Diphtheria; Hepatitis B | interventions — diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine

ARMS (2):
- INFANRIX HEXA 6-10-14 GROUP (Experimental): Healthy male or female subjects, aged between and including 6 and 10 weeks of age at the time of first vaccination, who received 3 doses of Infanrix hexa™ vaccine at 6, 10 and 14 weeks of age, administered intramuscularly in the right side of the thigh.
  Interventions: Biological: Infanrix hexa™
- INFANRIX HEXA 2-4-6 GROUP (Active Comparator): Healthy male or female subjects, aged between and including 6 and 10 weeks of age at the time of first vaccination, who received 3 doses of Infanrix hexa™ vaccine at 2, 4 and 6 months of age, administered intramuscularly in the right side of the thigh.
  Interventions: Biological: Infanrix hexa™

INTERVENTIONS:
Biological: Infanrix hexa™ — Intramuscular, three doses
  Other Names: DTPa-HBV-IPV/Hib

SUMMARY:
This study evaluates the immunogenicity and safety of Infanrix hexa™ (DTPa-HBV-IPV/Hib) when administered as a primary vaccination course to Indian infants according to a 6-10-14 weeks or a 2-4-6 months schedule.

ELIGIBILITY:
Inclusion Criteria:

All subjects must satisfy ALL the following criteria at study entry:

* A male or female between, and including, 6 and 10 weeks of age at the time of the first vaccination
* Documented administration of a hepatitis B vaccine dose at birth
* Subjects who the investigator believes that their parent(s)/legally acceptable representative(s) [LAR(s)] can and will comply with the requirements of the protocol
* Written informed consent obtained from the parent(s)/LAR(s) of the subject
* Healthy subjects as established by medical history and clinical examination before entering into the study
* Born after a gestation period of at least 36 weeks

Exclusion Criteria:

The following criteria should be checked at the time of study entry. If ANYexclusion criterion applies, the subject must not be included in the study:

* Child in care
* Use of any investigational or non-registered product other than the study vaccines within 30 days preceding the first dose, or planned use during the study period
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose
* Administration of a vaccine not foreseen by the study protocol, within 30 days prior to the first study visit, or planned administration during the study period, with the exception of oral human rotavirus (HRV) vaccination which is allowed at any time during the study
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product
* Evidence of previous diphtheria, tetanus, pertussis, hepatitis B, poliomyelitis and Haemophilus influenzae type b (Hib) vaccination or disease, with the exception of a birth dose of hepatitis B vaccine and oral poliovirus vaccine (OPV) as per local standard of care
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination
* Family history of congenital or hereditary immunodeficiency
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine
* Major congenital defects or serious chronic illness
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period
* Acute disease and/or fever at the time of enrolment

Ages: 6 Weeks to 10 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 224 (Actual)
Dates: Start 2012-04-16 (Actual); Primary Completion 2013-02-25 (Actual); Study Completion 2013-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- India (3):
  - GSK Investigational Site, Belgaun
  - GSK Investigational Site, Chennai
  - GSK Investigational Site, Pune

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=4632

REFERENCES:
- [Background] Lalwani SK, Agarkhedkar S, Sundaram B, Mahantashetti NS, Malshe N, Agarkhedkar S, Van Der Meeren O, Mehta S, Karkada N, Han HH, Mesaros N. Immunogenicity and safety of 3-dose primary vaccination with combined DTPa-HBV-IPV/Hib in Indian infants. Hum Vaccin Immunother. 2017 Jan 2;13(1):120-127. doi: 10.1080/21645515.2016.1225639. Epub 2016 Sep 15. PMID 27629913
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 111157 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111157 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111157 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111157 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111157 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111157 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Period: Overall Study
Arm/Group | Infanrix Hexa 6-10-14 Group | Infanrix Hexa 2-4-6 Group
Started | 112 | 112
Completed | 111 | 112
Not Completed | 1 | 0
Not completed — Migrated/moved from study area | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infanrix Hexa 6-10-14 Group | Infanrix Hexa 2-4-6 Group | Total
Number analyzed (Participants) | 112 | 112 | 224
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 6.7 (1.04) | 6.8 (1.13) | 6.75 (1.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 52 | 104
  Male | 60 | 60 | 120
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian-Central/South Asian heritage | 112 | 112 | 224

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroprotected Subjects Against Diphteria (D) and Tetanus (T) Antigens
Description: A seroprotected subject was defined as a vaccinated subject with anti-D and anti-T antibody concentration greater than or equal to (≥) 0.1 international units per milliliter (IU/mL).
Time Frame: One month post Dose 3 (Month 3 or Month 5)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, including all evaluable subjects for whom data was available for the considered timepoint and assay assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa 6-10-14 Group | Infanrix Hexa 2-4-6 Group
Number analyzed (Participants) | 105 | 106
Participants
  Anti-D | 105 | 106
  Anti-T | 105 | 106

2. Primary Outcome: Number of Seroprotected Subjects Against Hepatitis B (HBs)
Description: A seroprotected subject was defined as a vaccinated subject with anti-HBS antibody concentration ≥ 10 milli-international units per milliliter (mIU/mL).
Time Frame: One month post Dose 3 (Month 3 or Month 5)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa 6-10-14 Group | Infanrix Hexa 2-4-6 Group
Number analyzed (Participants) | 101 | 105
Participants | 101 | 104

3. Primary Outcome: Number of Seroprotected Subjects Against Poliovirus (Polio) Types 1,2,3 Antigens
Description: A seroprotected subject was defined as a subject with anti-Poliovirus 1,2 and 3 antibody titers ≥ 8 effective dose, for 50% of people receiving the vaccine (ED50).
Time Frame: One month post Dose 3 (Month 3 or Month 5)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa 6-10-14 Group | Infanrix Hexa 2-4-6 Group
Number analyzed (Participants) | 99 | 99
Participants
  Anti-Polio 1 | 99 | 99
  Anti-Polio 2: number analyzed (Participants) | 77 | 88
  Anti-Polio 2 | 77 | 88
  Anti-Polio 3: number analyzed (Participants) | 74 | 79
  Anti-Polio 3 | 73 | 79

4. Primary Outcome: Number of Seroprotected Subjects Against Polyribosyl-ribitol Phosphate (PRP) Antigens
Description: A seroprotected subject was defined as a subject with anti-PRP antibody concentration ≥ 0.15 micrograms per milliliter (µg/mL).
Time Frame: One month post Dose 3 (Month 3 or Month 5)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa 6-10-14 Group | Infanrix Hexa 2-4-6 Group
Number analyzed (Participants) | 105 | 106
Participants | 104 | 105

5. Primary Outcome: Number of Subjects With Vaccine Response for Pertussis Toxoid (PT), Filamentous Haemagglutinin (FHA) and Pertactin (PRN)
Description: Vaccine response was defined as : For initially seronegative subjects (S-), antibody concentration ≥ 5 enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/mL) at 1 month after the third dose; For initially seropositive subjects (S+): antibody concentration at 1 month after the third dose ≥ 1 fold increase in the pre-vaccination antibody concentration.
Time Frame: One month post Dose 3 (Month 3 or Month 5)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, including all evaluable subjects for whom data was available for the considered timepoint and assay assessed and for whom pre-vaccination data was available for the considered assay.
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa 6-10-14 Group | Infanrix Hexa 2-4-6 Group
Number analyzed (Participants) | 89 | 90
Participants
  Anti-PT, S-: number analyzed (Participants) | 61 | 67
  Anti-PT, S- | 61 | 67
  Anti-PT, S+: number analyzed (Participants) | 44 | 37
  Anti-PT, S+ | 44 | 36
  Anti-FHA, S-: number analyzed (Participants) | 12 | 12
  Anti-FHA, S- | 12 | 12
  Anti-FHA, S+ | 86 | 88
  Anti-PRN, S-: number analyzed (Participants) | 86 | 89
  Anti-PRN, S- | 86 | 89
  Anti-PRN, S+: number analyzed (Participants) | 19 | 15
  Anti-PRN, S+ | 18 | 14

6. Secondary Outcome: Anti-D and Anti-T Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in international units per milliliter (IU/mL).
Time Frame: One month post Dose 3 (Month 3 or Month 5)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Infanrix Hexa 6-10-14 Group | Infanrix Hexa 2-4-6 Group
Number analyzed (Participants) | 105 | 106
IU/mL
  Anti-D | 2.334 [2.049 to 2.659] | 3.726 [3.26 to 4.258]
  Anti-T | 3.307 [2.925 to 3.739] | 4.904 [4.378 to 5.493]

7. Secondary Outcome: Anti-HBs Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in milli-international units per milliliter (mIU/mL).
Time Frame: One month post Dose 3 (Month 3 or Month 5)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Infanrix Hexa 6-10-14 Group | Infanrix Hexa 2-4-6 Group
Number analyzed (Participants) | 101 | 105
mIU/mL | 1695.7 [1395.2 to 2060.9] | 3314.5 [2645.2 to 4153.1]

8. Secondary Outcome: Anti-Polio Types 1, 2, 3 Antibody Titers
Description: Antibody titers were presented as geometric mean titers (GMTs).
Time Frame: One month post Dose 3 (Month 3 or Month 5)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Infanrix Hexa 6-10-14 Group | Infanrix Hexa 2-4-6 Group
Number analyzed (Participants) | 99 | 99
Titers
  Anti-Polio 1 | 884.3 [666.6 to 1173.1] | 1799.2 [1429 to 2265.5]
  Anti-Polio 2: number analyzed (Participants) | 77 | 88
  Anti-Polio 2 | 840.2 [616.9 to 1144.2] | 2138.7 [1658.1 to 2758.7]
  Anti-Polio 3: number analyzed (Participants) | 74 | 79
  Anti-Polio 3 | 923.7 [691.9 to 1233.2] | 2245.5 [1866.1 to 2702.1]

9. Secondary Outcome: Anti-PRP Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in µg/mL.
Time Frame: One month post Dose 3 (Month 3 or Month 5)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Infanrix Hexa 6-10-14 Group | Infanrix Hexa 2-4-6 Group
Number analyzed (Participants) | 105 | 106
µg/mL | 2.697 [2.176 to 3.343] | 5.404 [4.168 to 7.006]

10. Secondary Outcome: Anti-PT, Anti-FHA and Anti-PRN Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in EL.U/mL.
Time Frame: One month post Dose 3 (Month 3 or Month 5)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Infanrix Hexa 6-10-14 Group | Infanrix Hexa 2-4-6 Group
Number analyzed (Participants) | 105 | 106
EL.U/mL
  Anti-PT | 107.3 [96.6 to 119.1] | 108.2 [97.4 to 120.2]
  Anti-FHA | 293.7 [259.4 to 332.6] | 369.3 [335.5 to 406.5]
  Anti-PRN | 224.4 [194.2 to 259.3] | 243.6 [213.2 to 278.4]

11. Secondary Outcome: Number of Seropositive Subjects for Anti-PT, Anti-FHA and Anti-PRN
Description: A seropositive subject was defined as a subject with anti-PT, anti-FHA and anti-PRN antibody concentrations ≥ 5 EL.U/mL.
Time Frame: One month post Dose 3 (Month 3 or Month 5)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa 6-10-14 Group | Infanrix Hexa 2-4-6 Group
Number analyzed (Participants) | 105 | 106
Participants
  Anti-PT | 105 | 106
  Anti-FHA | 105 | 106
  Anti-PRN | 105 | 106

12. Secondary Outcome: Number of Seroprotected Subjects Against Polio Type 1, 2 and 3 Antigens
Description: A seroprotected subject was defined as a subject with anti-Polio type 1, 2 and 3 antibody titers ≥ 8 effective dose, for 50% of people receiving the vaccine (ED50).
Time Frame: At Month 0
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa 6-10-14 Group | Infanrix Hexa 2-4-6 Group
Number analyzed (Participants) | 97 | 102
Participants
  Anti-Polio 1 | 71 | 70
  Anti-Polio 2: number analyzed (Participants) | 56 | 55
  Anti-Polio 2 | 38 | 42
  Anti-Polio 3: number analyzed (Participants) | 88 | 91
  Anti-Polio 3 | 23 | 30

13. Secondary Outcome: Number of Seropositive Subjects for Anti-PT, Anti-FHA and Anti-PRN
Description: A seropositive subject was defined as a subject with anti-PT, anti-FHA and anti-PRN antibody concentrations ≥ 5 EL.U/mL.
Time Frame: At Month 0
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa 6-10-14 Group | Infanrix Hexa 2-4-6 Group
Number analyzed (Participants) | 105 | 104
Participants
  Anti-PT | 44 | 37
  Anti-FHA: number analyzed (Participants) | 101 | 102
  Anti-FHA | 89 | 90
  Anti-PRN | 19 | 15

14. Secondary Outcome: Number of Seroprotected Subjects Against Anti-HBs Antigens
Description: A seroprotected subject was defined as a subject with anti-HBs antibody concentrations ≥ 10 mIU/mL.
Time Frame: At Month 0
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa 6-10-14 Group | Infanrix Hexa 2-4-6 Group
Number analyzed (Participants) | 80 | 81
Participants | 14 | 13

15. Secondary Outcome: Anti-Polio Types 1, 2 and 3 Antibody Titers
Description: Antibody titers were presented as geometric mean titers (GMTs).
Time Frame: At Month 0
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Infanrix Hexa 6-10-14 Group | Infanrix Hexa 2-4-6 Group
Number analyzed (Participants) | 97 | 102
Titers
  Anti-Polio 1 | 53.5 [33.5 to 85.3] | 31.9 [21.5 to 47.2]
  Anti-Polio 2: number analyzed (Participants) | 56 | 55
  Anti-Polio 2 | 32.5 [19.2 to 55] | 36.2 [22.2 to 59]
  Anti-Polio 3: number analyzed (Participants) | 88 | 91
  Anti-Polio 3 | 8 [5.9 to 10.8] | 11.9 [8.3 to 17]

16. Secondary Outcome: Anti-PT, Anti-FHA and Anti-PRN Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in EL.U/mL.
Time Frame: At Month 0
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Infanrix Hexa 6-10-14 Group | Infanrix Hexa 2-4-6 Group
Number analyzed (Participants) | 105 | 104
EL.U/mL
  Anti-PT | 5 [4.2 to 6] | 4.6 [3.8 to 5.6]
  Anti-FHA: number analyzed (Participants) | 101 | 102
  Anti-FHA | 18.7 [15 to 23.3] | 20.1 [16.1 to 25.2]
  Anti-PRN | 3.4 [2.9 to 3.9] | 3.2 [2.8 to 3.7]

17. Secondary Outcome: Anti-HBs Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in mIU/mL.
Time Frame: At Month 0
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Infanrix Hexa 6-10-14 Group | Infanrix Hexa 2-4-6 Group
Number analyzed (Participants) | 80 | 81
mIU/mL | 5.9 [4.2 to 8.3] | 5.6 [4.1 to 7.7]

18. Secondary Outcome: Number of Subjects With Any Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = incidence of any particular symptom regardless of intensity grade.
Time Frame: During the 4-day (Days 0-3) post-vaccination period after each dose and across doses: Up to Month 2 (Infanrix Hexa 6-10-14 Group) or Month 4 (Infanrix Hexa 2-4-6 Group)
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects who received at least one dose of the study vaccine, for whom data were available and who had the symptoms sheet filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa 6-10-14 Group | Infanrix Hexa 2-4-6 Group
Number analyzed (Participants) | 111 | 112
Participants
  Any Pain, Dose 1 | 23 | 11
  Any Redness, Dose 1 | 3 | 1
  Any Swelling, Dose 1 | 7 | 4
  Any Pain, Dose 2 | 13 | 3
  Any Redness, Dose 2 | 0 | 1
  Any Swelling, Dose 2 | 2 | 2
  Any Pain, Dose 3 | 10 | 6
  Any Redness, Dose 3 | 3 | 0
  Any Swelling, Dose 3 | 2 | 3
  Any Pain, Across doses | 28 | 15
  Any Swelling, Across doses | 6 | 2
  Any Redness, Across doses | 8 | 9

19. Secondary Outcome: Number of Subjects With Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, irritability/fussiness, loss of appetite and temperature [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)]. Any = incidence of any particular symptom regardless of intensity grade or relationship to study vaccination.
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Groups:
- Infanrix Hexa 6-10-14 Group: Healthy male or female subjects, aged between and including 6 and 10 weeks of age at the time of first vaccination, who received 3 doses of Infanrix hexa vaccine at 6, 10 and 14 weeks of age, administered intramuscularly in the right side of the thigh.
- Infanrix Hexa 2-4-6 Group: Healthy male or female subjects, aged between and including 6 and 10 weeks of age at the time of first vaccination, who received 3 doses of Infanrix hexa vaccine at 2, 4 and 6 months of age, administered intramuscularly in the right side of the thigh.
Arm/Group | Infanrix Hexa 6-10-14 Group | Infanrix Hexa 2-4-6 Group
Number analyzed (Participants) | 111 | 112
Participants
  Any Drowsiness, Dose 1 | 0 | 2
  Any Irritability/fussiness, Dose 1 | 8 | 5
  Any Loss of appetite, Dose 1 | 1 | 3
  Any Temperature/(Axillary), Dose 1 | 10 | 7
  Any Drowsiness, Dose 2 | 0 | 0
  Any Irritability/fussiness, Dose 2 | 2 | 5
  Any Loss of appetite, Dose 2 | 0 | 1
  Any Temperature/(Axillary), Dose 2 | 5 | 7
  Any Drowsiness, Dose 3 | 0 | 0
  Any Irritability/fussiness, Dose 3 | 3 | 3
  Any Loss of appetite, Dose 3 | 1 | 1
  Any Temperature/(Axillary), Dose 3 | 3 | 6
  Any Drowsiness, Across doses | 0 | 2
  Any Irritability/fussiness, Across doses | 13 | 10
  Any Loss of appetite, Across doses | 2 | 5
  Any Temperature/(Axillary), Across doses | 17 | 17

20. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-day (Days 0-30) post-vaccination period: Up to Month 3 (Infanrix Hexa 6-10-14 Group) or Month 5 (Infanrix Hexa 2-4-6 Group)
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects who received at least one dose of the study vaccine and for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa 6-10-14 Group | Infanrix Hexa 2-4-6 Group
Number analyzed (Participants) | 112 | 112
Participants | 40 | 25

21. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (from Month 0 up to Month 3 (Infanrix Hexa 6-10-14 Group) or Month 5 (Infanrix Hexa 2-4-6 Group))
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix Hexa 6-10-14 Group | Infanrix Hexa 2-4-6 Group
Number analyzed (Participants) | 112 | 112
Participants | 2 | 3

ADVERSE EVENTS:
Time Frame: Solicited symptoms: during the 4-day (Days 0-3) post-vaccination period. Unsolicited AEs: during the 31-day (Days 0-30) post-vaccination period. SAEs: during the entire study period (from Month 0 to Month 3 or Month 5).
Arm/Group | Infanrix Hexa 6-10-14 Group | Infanrix Hexa 2-4-6 Group
All-Cause Mortality (participants affected / at risk) | 0/112 | 0/112
Serious Adverse Events (participants affected / at risk) | 2/112 | 3/112
Other Adverse Events (participants affected / at risk) | 45/112 | 36/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infanrix Hexa 6-10-14 Group (N=112) | Infanrix Hexa 2-4-6 Group (N=112)
Lower respiratory tract infection (Infections and infestations) | 0 | 2
Bronchiolitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infanrix Hexa 6-10-14 Group (N=112) | Infanrix Hexa 2-4-6 Group (N=112)
Erythema (Skin and subcutaneous tissue disorders) | 6 (6) | 2 (2)
Irritability (Psychiatric disorders) | 13 (13) | 10 (13)
Pain (General disorders) | 28 (46) | 15 (20)
Pyrexia (General disorders) | 18 (19) | 17 (20)
Rhinitis (Infections and infestations) | 4 (5) | 6 (6)
Swelling (General disorders) | 8 (11) | 9 (9)
Upper respiratory tract infection (Infections and infestations) | 18 (23) | 11 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.